CLINICAL TRIAL: NCT03631563
Title: Comparing ATG-Fresenius vs Thymoglobulin for the Prevention of Graft-versus-host Disease in the Setting of Haplo-identical Hematopoietic Stem Cell Transplantation
Brief Title: ATG-F VS ATG for the Prevention of GVHD
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fujian Medical University (Other)
Responsible Party: Principal Investigator, Ting YANG, Prof.M.D.Ph.D, Fujian Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ATG-F VS ATG-01
Record Dates: First submitted 2018-08-13; First posted 2018-08-15 (Actual); Last update posted 2018-08-15 (Actual); Status verified 2018-08

CONDITIONS: GVHD in the Setting of Haplo-HSCT
MeSH Terms: interventions — Immunosuppressive Agents

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Experimental): ATG-F treated
  Interventions: Drug: Immunosuppressive Agent
- Arm 2 (Active Comparator): ATG treated
  Interventions: Drug: Immunosuppressive Agent

INTERVENTIONS:
Drug: Immunosuppressive Agent — ATG-Fresenius versus ATG

SUMMARY:
Anti-thymocyte globulin (ATG) preparative regimen in the setting of haploidentical stem cell transplantation (haplo-HSCT) is vital for inducing immune tolerance.The study aims to compare the efficacy and safety of ATG-F vs ATG, incorporated into the preparative regimens for haplo-identical transplants.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent
* Aged <65 years
* Patients undergoing Haplo-identical hematopoietic stem cell transplantation.
* Cardiac: Left ventricular ejection fraction ≥ 50%
* Adequate renal and hepatic function
* Performance status: Karnofsky ≥ 70%

Exclusion Criteria:

* Pregnant or lactating females.
* Any co-morbidity precluding the administration of ATG or ATG-F.

Max Age: 65 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2013-03-01 (Actual); Primary Completion 2018-12-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
incidence of GVHD | 1 year

SECONDARY OUTCOMES:
leukemia-free survival | 1 year
treatment-related mortality | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Fujian Medical University Union Hospital, Fuzhou, Fujian, China